CLINICAL TRIAL: NCT00275236
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, Two-arm, Parallel-group, Sleep Lab Trial to Investigate the Efficacy and Safety of Transdermal Rotigotine in Subjects With Idiopathic Restless Legs Syndrome
Brief Title: A Sleep Lab Trial to Investigate the Efficacy and Safety of Transdermal Rotigotine in Subjects With Idiopathic Restless Legs Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0794; 2005-002814-39 (EudraCT Number)
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Restless Legs Syndrome
Keywords: Idiopthic Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — rotigotine

INTERVENTIONS:
Drug: Rotigotine

SUMMARY:
The objective of this trial is to demonstrate that rotigotine (SPM 936) is effective in subjects with idiopathic RLS based on the PLMI (Periodic Limb Movements Index)(PLMs/total time in bed) as measured by polysomnography (PSG). The primary variable is the reduction of PLMI at the end of the Maintenance Period compared to Baseline. PLMI data will be obtained from PSGs.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic RLS

Exclusion Criteria:

* secondary RLS
* history of sleep disturbances
* symptomatic orthostatic hypotension

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-11; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Efficacy is assessed by reduction of Periodic Limb Movement Index, which will be obtained from polysomnographic measurements.

SECONDARY OUTCOMES:
Changes in Periodic Limb Movement Arousal Index, Sleep efficiency, International RLS sum score, Clinical Global Impression Item 1.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- Schwarz BioSciences, Monheim, Germany

REFERENCES:
- [Result] Oertel WH, Benes H, Garcia-Borreguero D, Hogl B, Poewe W, Montagna P, Ferini-Strambi L, Sixel-Doring F, Trenkwalder C, Partinen M, Saletu B, Polo O, Fichtner A, Schollmayer E, Kohnen R, Cassel W, Penzel T, Stiasny-Kolster K. Rotigotine transdermal patch in moderate to severe idiopathic restless legs syndrome: a randomized, placebo-controlled polysomnographic study. Sleep Med. 2010 Oct;11(9):848-56. doi: 10.1016/j.sleep.2010.02.014. Epub 2010 Sep 1. PMID 20813583